CLINICAL TRIAL: NCT03307811
Title: Endoscopic Ultrasound Guided Liver Biopsy Using a 22 Gauge Fine Needle Biopsy Needle.
Brief Title: Endoscopic Ultrasound Guided Liver Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1055744
Record Dates: First submitted 2017-07-17; First posted 2017-10-12 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Hepatic Cancer; Hepatic Neoplasm; Hepatic Carcinoma
Keywords: liver; biopsy; hepatic; EUS; fine needle biopsy
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 22 gauge needle liver biopsy (Experimental): EUS-LB will be performed using a 22 g FNB needle. Specimens obtained from each pass will be placed in a separate biopsy jar. If the third pass does not result in sufficient diagnostic material, a 19 G will be used. A maximum of 3 passes will be made using the alternate needle. The total number of passes with the 22 G needle and the 19 G needle is 6. Data will be collected about the procedure and the performance of the needles for each procedure.
  Interventions: Other: 22 gauge needle liver biopsy

INTERVENTIONS:
Other: 22 gauge needle liver biopsy — EUS will be performed. Specimens obtained from each pass will be placed in a separate biopsy jar. If the third pass does not result in sufficient diagnostic material, a 19 G will be used. A maximum of 3 passes will be made using the alternate needle. The total number of passes with the 22 G needle and the 19 G needle is 6. Data will be collected about the procedure and the performance of the needles for each procedure.

SUMMARY:
This is a prospective study to determine the optimal technique for obtaining liver tissue with a smaller caliber (22 gauge) needle and whether a good core biopsy can be obtained without the use of suction and secondly to determine the diagnostic yield and safety of 22 g Fine Needle Biopsy needle for liver biopsy.

DETAILED DESCRIPTION:
Liver biopsy (LB) has historically been performed by percutaneous route without image guidance (blind biopsy). However, in the last several years there has been more reliance on image guidance ultrasound-guided (USG) or computed tomography (CT) to direct the needle into the liver with the hope of limiting complications. Other ways of performing liver biopsy are transjugular fluoroscopy guided approach when percutaneous route is deemed not safe because of coagulopathy or ascites. Surgical LB (either laparoscopic or open) is yet another way of obtaining liver tissue.

Endoscopic ultrasound guided liver biopsy (EUS-LB) is proposed as a newer method that may offer several potential advantages over existing techniques for attaining liver tissue. It can be performed in an outpatient setting and offers the comfort of sedation and analgesia. Endoscopic Ultrasound (EUS) provides high resolution images of left lobe of the liver and a good portion of the right lobe of the liver. This coupled with Doppler capability the biopsy needle can be safely directed into the liver for sampling under real time image guidance. Intervening structures such as pleura, bowel loops and gallbladder can be easily seen by EUS and thus avoided that further decreases the risk of adverse events. It has been recognized that sampling error can lead to diagnostic inaccuracy of a biopsy from a single site. As compared to USG or CT scan the EUS allows easy and safe biopsy of both left and right lobes of the liver during same setting, potentially addressing concerns about sampling error.

The cost of the endoscopic procedure is the main expense of EUS-LB. Thus this approach is best used for patients requiring EUS for evaluation of elevated liver tests. If no obstructive lesion is identified by EUS that will require endoscopic retrograde cholangiopancreatography (ERCP) then it would cost-effective to perform EUS-LB during the same setting without much additional time and risks. This approach can spare the patient the additional discomfort and expense of a second dedicated LB procedure by any of the other available techniques (percutaneous, transjugular etc.). In such setting the equipment costs for the EUS-LB will mainly include only the Fine Needle Biopsy (FNB) needle, which is similar in expense to the cost of needles for the transjugular or percutaneous approach.

The traditionally used transcutaneous LB needle is 16 gauge (G) while largest EUS biopsy needle is 19 G. The smaller size of the needle is expected to decrease the complications rate (mainly pain and bleeding) even further. Many studies using a 19 G Tru-cut biopsy or Fine Needle Aspiration (FNA) needle to acquire liver tissue have obtained specimens adequate for histologic diagnosis but there has been a wide range of specimen adequacy (19-100%). The 19 G Tru-cut biopsy needle has been associated with several technical difficulties that could reflect negatively on tissue adequacy.

While it is easy and straight forward to biopsy the left lobe of the liver with any EUS needle. The 19 G needle is a large bore needle for EUS use and it is sometimes difficult to attain an adequate position for biopsy specially in duodenum where scope is torqued and this is the only area of access to right lobe.

In this study the investigators will use a 22 G needle. Smaller caliber of the needle would not only make it technically easier to access right lobe of the liver through the duodenum, it is also expected to decrease the risks further due to smaller size. Also, the 22 G EUS-FNB needle has three cutting points at the cutting edge of the needle that provide stability at puncture while the high quality, fully formed heels are designed to maximize tissue capture and minimize fragmentation, that would result in attaining a good histological specimen, a main stay for liver biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. All patients referred to Florida Hospital Endoscopy Unit for assessment of elevated liver tests with EUS and are found to have no obstructive lesion to explain elevation of liver tests and will not require ERCP.
2. Age ≥ 19 years
3. Willing to provide informed consent verbal or written.

Exclusion Criteria:

1. Age <19 years
2. Unable to safely undergo EUS for any reason
3. Coagulopathy (INR >1.6, Thrombocytopenia with platelet count <50,000/ml) for subjects on anti-coagulation therapy.
4. Unwilling or cognitively unable to provide informed consent verbal or written.
5. Pregnancy (confirmed with Standard of Care urine pregnancy test for all women with child-bearing potential only)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-06-19 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic adequacy of the liver biopsy specimen | Sample obtained during EUS-guided liver biopsy.
  Determine the diagnostic adequacy of the liver biopsy specimen by obtaining a histological specimen using a smaller (22 G) caliber needle. Diagnostic adequacy is defined as a sample that provides definitive pathological diagnosis (yes, no).

SECONDARY OUTCOMES:
Visible core | Sample obtained during EUS-guided liver biopsy.
  The sample will have a visible core (yes/no).
Suction | Sample obtained during EUS-guided liver biopsy.
  Sample was obtained using suction (yes/no).
Number of passes required histological samples | Time of Liver biopsy
  Assessing the median number of passes required to obtain diagnostically adequate histological samples histological samples
Technical failure | Time of Liver biopsy
  Was there a technical failure (yes/no).
Complications/Bleeding | 1 month
  Assessing subjects for post-procedural complications via follow up phone calls. Bleeding (yes/no).
Complications/Pain | 1 month
  Assessing subjects for post-procedural complications via follow up phone calls. Pain (yes/no).
Complications/Infection | 1 Month
  Assessing subjects for post-procedural complications via follow up phone calls. Infection (yes/no).

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hasan, MD, Principal Investigator — Florida Hospital - Center for Interventional Endoscopy
Locations (1):
- Center for Interventional Endoscopy - Florida Hospital, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the individual participant data with other researchers.

REFERENCES:
- [Background] Rockey DC, Caldwell SH, Goodman ZD, Nelson RC, Smith AD; American Association for the Study of Liver Diseases. Liver biopsy. Hepatology. 2009 Mar;49(3):1017-44. doi: 10.1002/hep.22742. No abstract available. PMID 19243014
- [Background] Kalambokis G, Manousou P, Vibhakorn S, Marelli L, Cholongitas E, Senzolo M, Patch D, Burroughs AK. Transjugular liver biopsy--indications, adequacy, quality of specimens, and complications--a systematic review. J Hepatol. 2007 Aug;47(2):284-94. doi: 10.1016/j.jhep.2007.05.001. Epub 2007 May 24. PMID 17561303
- [Background] Mathew A. EUS-guided routine liver biopsy in selected patients. Am J Gastroenterol. 2007 Oct;102(10):2354-5. doi: 10.1111/j.1572-0241.2007.01353_7.x. No abstract available. PMID 17897349
- [Background] Gleeson FC, Clayton AC, Zhang L, Clain JE, Gores GJ, Rajan E, Smyrk TC, Topazian MD, Wang KK, Wiersema MJ, Levy MJ. Adequacy of endoscopic ultrasound core needle biopsy specimen of nonmalignant hepatic parenchymal disease. Clin Gastroenterol Hepatol. 2008 Dec;6(12):1437-40. doi: 10.1016/j.cgh.2008.07.015. Epub 2008 Jul 26. PMID 19081532
- [Background] Dewitt J, McGreevy K, Cummings O, Sherman S, Leblanc JK, McHenry L, Al-Haddad M, Chalasani N. Initial experience with EUS-guided Tru-cut biopsy of benign liver disease. Gastrointest Endosc. 2009 Mar;69(3 Pt 1):535-42. doi: 10.1016/j.gie.2008.09.056. PMID 19231495
- [Background] Stavropoulos SN, Im GY, Jlayer Z, Harris MD, Pitea TC, Turi GK, Malet PF, Friedel DM, Grendell JH. High yield of same-session EUS-guided liver biopsy by 19-gauge FNA needle in patients undergoing EUS to exclude biliary obstruction. Gastrointest Endosc. 2012 Feb;75(2):310-8. doi: 10.1016/j.gie.2011.09.043. PMID 22248599
- [Background] Nakai Y, Samarasena JB, Iwashita T, Park DH, Lee JG, Hu KQ, Chang KJ. Autoimmune hepatitis diagnosed by endoscopic ultrasound-guided liver biopsy using a new 19-gauge histology needle. Endoscopy. 2012;44 Suppl 2 UCTN:E67-8. doi: 10.1055/s-0031-1291567. Epub 2012 Mar 6. No abstract available. PMID 22396285
- [Background] Maharaj B, Maharaj RJ, Leary WP, Cooppan RM, Naran AD, Pirie D, Pudifin DJ. Sampling variability and its influence on the diagnostic yield of percutaneous needle biopsy of the liver. Lancet. 1986 Mar 8;1(8480):523-5. doi: 10.1016/s0140-6736(86)90883-4. PMID 2869260
- [Background] Diehl DL, Johal AS, Khara HS, Stavropoulos SN, Al-Haddad M, Ramesh J, Varadarajulu S, Aslanian H, Gordon SR, Shieh FK, Pineda-Bonilla JJ, Dunkelberger T, Gondim DD, Chen EZ. Endoscopic ultrasound-guided liver biopsy: a multicenter experience. Endosc Int Open. 2015 Jun;3(3):E210-5. doi: 10.1055/s-0034-1391412. Epub 2015 Feb 27. PMID 26171433